CLINICAL TRIAL: NCT05305222
Title: A Study in Healthy Japanese and Caucasian Subjects to Assess the Pharmacokinetics, Safety and Tolerability After a Single Dose of Risankizumab
Brief Title: A Study in Healthy Japanese and Caucasian Subjects to Assess the Pharmacokinetics, Safety and Tolerability of Risankizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M16-533
Record Dates: First submitted 2022-03-23; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Risankizumab; Skyrizi
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Japanese Participants Receiving Risankizumab (Experimental): Participants will receive single dose of risankizumab.
  Interventions: Drug: Risankizumab
- Japanese Participants Receiving Placebo (Experimental): Participants will receive single dose of placebo.
  Interventions: Drug: Placebo
- Caucasian Participants Receiving Risankizumab (Experimental): Participants will receive single dose of risankizumab.
  Interventions: Drug: Risankizumab
- Caucasian Participants Receiving Placebo (Experimental): Participants will receive single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risankizumab — Intravenous (IV) Infusion
  Other Names: SKYRIZI; ABBV-066
  Arms: Caucasian Participants Receiving Risankizumab; Japanese Participants Receiving Risankizumab
Drug: Placebo — Intravenous (IV) Infusion
  Arms: Caucasian Participants Receiving Placebo; Japanese Participants Receiving Placebo

SUMMARY:
The main objective of this study is to assess the pharmacokinetics, safety, tolerability and immunogenicity following a single intravenous (IV) infusion of risankizumab in healthy Japanese and Caucasian participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be first or second generation Japanese of full parentage residing outside of Japan for less than 10 years. First generation participants will have been born to two parents and four grandparents also born in Japan of full Japanese descent. Second generation participants born outside of Japan must have two parents and four grandparents born in Japan of full Japanese descent. All participants must maintain a typical Japanese lifestyle, including consuming a typical Japanese diet or participants must be Caucasian and not of Hispanic ethnicity.
* Body Mass Index (BMI) is >= 18.5 and <= 29.9 kg/m2 (after rounding to the tenths decimal) at Screening. BMI is calculated as weight in kilograms (kg) divided by the square of height measured in meters (m).

Exclusion Criteria:

* Previous exposure to any anti-IL-12/23 or anti-IL-23 treatment.
* Any findings in the medical examination that are deviating from normal and judged as clinically relevant by the investigator.
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease judged as clinically relevant by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 137 days
  An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Plasma Concentration (Cmax) of Risankizumab | Up to approximately 137 days
  Maximum observed plasma concentration (Cmax) of Risankizumab.
Time to Cmax (Cmax) of Risankizumab | Up to approximately 137 days
  Tmax of Risankizumab.
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Last Measurable Concentration (AUCt) of Risankizumab | Up to approximately 137 days
  AUCt of Risankizumab.
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Infinity (AUCinf) of Risankizumab | Up to approximately 137 days
  AUCinf of Risankizumab.
Apparent Terminal Phase Elimination Rate Constant (β) of Risankizumab | Up to approximately 137 days
  Apparent terminal phase elimination rate constant (β) of Risankizumab.
Terminal Phase Elimination Half-life (t1/2) of Risankizumab | Up to approximately 137 days
  Terminal phase elimination half-life (t1/2) of Risankizumab.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Altasciences Clinical Los Angeles, Inc /ID# 164197, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No